CLINICAL TRIAL: NCT04567095
Title: A Cross-sectional Study Among Patients in Canada to Assess Awareness and Knowledge of the Fibristal Patient Alert Card
Brief Title: A Study to Evaluate Awareness and Knowledge of the Fibristal Additional Risk Minimization Measures Among Patients in Canada
Status: Withdrawn | Type: Observational
Why Stopped: This study was cancelled before any data collection due to business reasons.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: CMO-EPI-WH-0626
Record Dates: First submitted 2020-09-01; First posted 2020-09-28 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional, cross-sectional survey study to evaluate the effectiveness of the Additional Risk Minimization Measures for Fibristal among Patients in Canada.

DETAILED DESCRIPTION:
Data will be collected via web-based data capture and paper surveys depending on patient preference. The survey will be conducted in a single wave over 6 months. All data will be maintained in compliance with local regulations.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received Fibristal within 6 months of completing the survey.
* Patients who have provided permission to share their responses in aggregate with Health Canada.
* Patients who have provided informed consent for their participation in the survey.

Exclusion Criteria:

* Patients who participated in the cognitive pre-testing of the survey questionnaire to be used for the study.
* Patients who have been direct employees of Allergan, ICON, Health Canada, or Professional Targeted Marketing (PTM) within the past year.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The survey will endeavor to collect 150 completed patient surveys
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentages of patients with correct responses to the knowledge related questions based on the contents of the Fibristal Patient Alert Card. | 18 - 24 months
  Correct responses to knowledge-related questions (i.e, potential of fibristal to cause liver injury, signs and symptoms of liver problems, and what to do in case of signs and symptoms of liver problems.)

SECONDARY OUTCOMES:
Percentages of patients that recall recieving and using the Fibristal Patient Alert Card | 18 - 24 months
  Receipt and use of the Fibristal Patient Alert Card,
Percentage of patients that recall their HCPs' ordering of required liver function tests in accordance with the recommendations in the aRMM/CPM | 18 - 24 months
  Timing and frequency of liver testing conducted by the patients's HCP

CONTACTS AND LOCATIONS:
Overall Officials: Ahunna Ukah, Study Director — Allergan
Locations (1):
- Clinical Trials Registry Team, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Allergan will share de-identified patient-level data and study-level data including protocols and clinical study reports for phase 2 - 4 trials completed after 2008 that are registered to ClinicalTrials.gov or EudraCT, have received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published. To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes. More information can be found on http://www.allerganclinicaltrials.com/.
Supporting Information: Study Protocol, CSR
Time Frame: After having received regulatory approval in the United States and/or the European Union in a given indication and the primary manuscript from the trial has been published.
Access Criteria: To request access to the data, the researcher must sign a data use agreement and any shared data is to be used for non-commercial purposes.
URL: http://www.allerganclinicaltrials.com/